CLINICAL TRIAL: NCT00041899
Title: Pharmacokinetic Comparison of Two Preparations of the Selective Progesterone Receptor Modular CDB2914
Brief Title: Comparison of Blood Levels of Two Formulations of the Selective Hormone Receptor Modulator CDB-2914
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020219; 02-CH-0219
Record Dates: First submitted 2002-07-18; First posted 2002-07-19 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-03

CONDITIONS: Healthy
Keywords: Progesterone; Cortisol; Menstrual Cycle; Formulation; Endometrium; Estrogen
MeSH Terms: interventions — ulipristal

INTERVENTIONS:
Drug: CDB-2914
Drug: COB-2914

SUMMARY:
This study will compare blood levels of the drug CDB-2914 in healthy women receiving the compound in crystalline powder form with the blood levels of women receiving an identical dose of the drug in micronized form. Generally, absorption of compounds made into a crystalline powder is less than that of micronized compounds, in which the substance is processed into many similar-sized particles.

CDB-2914 is a manmade hormone similar to the hormones cortisol and progesterone. The National Institute of Child Health and Human Development is evaluating the ability of this drug to treat reproductive conditions. Institute studies have shown that CDB-2914 can increase the time to produce a mature egg in the ovary, and cause an early menstrual period, CDB-2914 might be used to treat fibroids and endometriosis pain. As part of its evaluation for these purposes, this study will determine if absorption of crystalline and micronized powder forms of CDB-2914 result in the same blood levels of the drug.

Women between 18 and 50 years of age who are in good health may be eligible for this study. Premenopausal women must not be pregnant (as determined by a urine pregnancy test) or breastfeeding and must practice birth control during the study. Candidates will be screened with a medical history, physical examination, and blood and urine tests. Women who use an IUD for contraception are advised to also use a barrier contraceptive (diaphragm or condom) the week after taking CDB-2914.

Participants will be admitted to the NIH Clinical Center inpatient service or the outpatient day hospital twice for pharmacokinetic studies (blood drawing to measure blood levels of CDB-2914 after a single dose of the drug). They will come to the Clinical Center at 7:00 a.m. and have a catheter (thin plastic tube) inserted into an arm vein for drawing blood for the first 24 hours of the study. Eight milliliters (about 2 teaspoons) of blood will be drawn 5 minutes and 1 minute before taking CDB-2914 (in either crystalline or micronized powder form) and then at the following times after taking the drug: 15, 30, 45, 60, 75, 90, 105, 120, 150 and 180 minutes (3 hours), and 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 hours (5 days).

Participants will take all their meals in the day hospital or ward during the first 26 hours of sampling. Inpatients will leave the hospital after the 24-hour blood draw and return as an outpatient on days 2 through 5. At the 48-hour time point, additional blood will be drawn to check blood counts and chemistries, and for liver and kidney function tests.

DETAILED DESCRIPTION:
In recent years, compounds that are structurally similar to the naturally occurring steroids have been examined for their ability to block or substitute for the action of the naturally occurring steroids. On occasion, these substances have both effects, depending on the tissue that is examined or on the physiology of the person receiving the agent. The development of these kinds of compounds, called selective hormone receptor modulators, may provide new treatments that are targeted to specific organs or tissues. One example of these compounds is the selective estrogen receptor modulator raloxifene, which blocks estrogen action at the uterus, and acts like estrogen at the bone, allowing its use in post-menopausal women as estrogen replacement therapy without requiring progesterone.

This study evaluates the progesterone receptor modulator CDB-2914. Earlier studies using single doses of this compound show that it can slow ovarian and uterine development during the menstrual cycle, and can induce menses, depending on when it is given during the menstrual cycle.

Many steroids have an improved bioavailability when given in a micronized formulation. Previous studies with CDB-2914 have used crystalline powder up to a dose of 200 mg. We wish to compare the pharmacokinetic profile of crystalline and micronized CDB-2914, 10 mg. The drug will be given as a single oral dose and blood will be drawn frequently over 12 hours and then daily for five days for measurement of the compound.

ELIGIBILITY:
INCLUSION CRITERIA:

General inclusion criteria:

Female gender--to evaluate effects in the target population for clinical trials.

In good health. Chronic medication use is acceptable except for glucocorticoid use. Other chronic medication use may be acceptable at discretion of the principal investigator. Interval use of over-the-counter drugs is acceptable but must be recorded.

Hemoglobin greater than 10 g/dL.

Willing and able to comply with study requirements.

Age 18 to 50.

Additional inclusion criteria for pre-menopausal women:

Using mechanical (condoms, diaphragms), abstinence, oral contraceptive, IUD or sterilization methods of contraception for the duration of the study. Because the effect of CDB-2914 on IUD efficacy is not known, women using this form of birth control will be advised to use barrier methods during the cycle(s) in which they participate.

Negative urine pregnancy test within one week of the first study. If the second study occurs in a subsequent cycle, the pregnancy test will be repeated.

EXCLUSION CRITERIA:

Significant abnormalities in the history, physical or laboratory examination

Pregnancy

Lactation

Use of oral, injectable or inhaled glucocorticoids or megesterol within the last year

Unexplained vaginal bleeding

History of malignancy within the past 5 years

Use of anti-epileptic agents

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 2002-05; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Batista MC, Cartledge TP, Zellmer AW, Merino MJ, Axiotis C, Loriaux DL, Nieman LK. Delayed endometrial maturation induced by daily administration of the antiprogestin RU 486: a potential new contraceptive strategy. Am J Obstet Gynecol. 1992 Jul;167(1):60-5. doi: 10.1016/s0002-9378(11)91627-5. PMID 1442957
- [Background] Cadepond F, Ulmann A, Baulieu EE. RU486 (mifepristone): mechanisms of action and clinical uses. Annu Rev Med. 1997;48:129-56. doi: 10.1146/annurev.med.48.1.129. PMID 9046951
- [Background] D'Argenio DZ, Schumitzky A. A program package for simulation and parameter estimation in pharmacokinetic systems. Comput Programs Biomed. 1979 Mar;9(2):115-34. doi: 10.1016/0010-468x(79)90025-4. PMID 761456